CLINICAL TRIAL: NCT06576427
Title: Selective Pulmonary-artery Intervention to Reduce Acute Right-heart tEnsion-II
Acronym: SPIRARE II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jupiter Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-02
Record Dates: First submitted 2024-04-18; First posted 2024-08-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Embolism
Keywords: Embolism and Thrombosis; Pulmonary Embolism; Embolism; Cardiovascular Diseases
MeSH Terms: conditions — Pulmonary Embolism; Embolism and Thrombosis; Embolism; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Vertex Pulmonary Embolectomy System (Experimental): Patients presenting with clinical signs and symptoms of acute PE and who meet the study criteria will be treated with the Vertex Pulmonary Embolectomy System
  Interventions: Device: Vertex Pulmonary Embolectomy System

INTERVENTIONS:
Device: Vertex Pulmonary Embolectomy System — Use of Vertex Pulmonary Embolectomy System to treat pulmonary embolism.

SUMMARY:
This study is a prospective, single-arm, multicenter study to evaluate the safety and effectiveness of the Vertex Pulmonary Embolectomy System in participants presenting with clinical signs and symptoms of acute pulmonary embolism.

DETAILED DESCRIPTION:
The study is a prospective, single-arm, multicenter study to evaluate the safety and effectiveness of the Vertex Pulmonary Embolectomy System in participants presenting with clinical signs and symptoms of acute pulmonary embolism.

The Vertex Pulmonary Embolectomy System is intended for the non-surgical removal of emboli and thrombi from blood vessels as a means for treating pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria

1. . Age ≥ 18 years < 80 years
2. Acute onset of symptoms < 14 days consistent with the presence of pulmonary embolism.
3. CTA evidence (site determined) of proximal PE (filling defect in at least one main or interlobar pulmonary artery)
4. RV/LV ratio of > 0.9 on CTA as assessed by investigator (site determined).
5. Systolic blood pressure ≥ 90 mmHg (initial SBP may be ≥ 80 mmHg if the pressure recovers to ≥ 90 mmHg with fluids)
6. Subject or subject's legally authorized representative (LAR) - applicable for US is willing and able to provide written informed consent prior to receiving any non-standard of care Clinical Investigation Plan-specific procedures
7. Subject is willing and able to comply with all Clinical Investigation Plan required follow-up visits

Exclusion Criteria

1. Thrombolytic use within 30 days of baseline CTA
2. Pulmonary hypertension with peak pulmonary artery pressure > 70 mmHg by right heart catheterization (site determined)
3. Vasopressor requirement after fluids to keep pressure ≥ 90 mmHg
4. Unstable heart rate > 130 beats per minute prior to procedure
5. FiO2 requirement > 40% or > 6 LPM to keep oxygen saturation > 90%
6. Hematocrit < 28%
7. Platelets < 100,000/μL
8. Serum baseline creatinine > 1.8 mg/dL
9. International normalized ratio (INR) > 3
10. Major trauma injury severity score (ISS) > 15 within the past 14 days
11. Presence of intracardiac lead in the right ventricle or right atrium placed <180 days prior to the index procedure
12. Cardiovascular or pulmonary surgery within last 30 days
13. Actively progressing cancer requiring chemotherapy
14. Known bleeding diathesis or coagulation disorder
15. Left bundle branch block
16. History of severe or chronic pulmonary arterial hypertension
17. History of chronic left heart disease with left ventricular ejection fraction ≤ 30%
18. History of decompensated heart failure
19. Patients on extracorporeal membrane oxygenation (ECMO)
20. History of underlying lung disease that is oxygen dependent
21. History of chest irradiation
22. History of heparin-induced thrombocytopenia (HIT)
23. Contraindication to systemic or therapeutic doses of heparin or anticoagulants
24. Known anaphylactic reaction to radiographic contrast agents that cannot be pretreated
25. Imaging evidence or other evidence that suggests, in the opinion of the Investigator, the Subject is not appropriate for mechanical thrombectomy intervention
26. Life expectancy of < 365 days, as determined by Investigator
27. Female who is pregnant or nursing
28. Current participation in another investigational drug or device treatment study
29. Inability to lay flat for procedure
30. Known presence of right-to-left cardiac shunt
31. History of Hemorrhagic or Ischemic Stroke, including Transient Ischemic Attack, within last 90 days
32. Current or history of chronic thromboembolic pulmonary hypertension (CTEPH) or chronic thromboembolic disease (CTED) diagnosis

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-02-04 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Reduction in Right ventricle (RV) / Left Ventricle (LV) ratio | From baseline to 48 hours or discharge
  Reduction in RV/LV ratio from baseline to 48 hours or discharge by (core lab assessed) CT angiography
Major Adverse Events, a composite of: | Within 48 hours of the procedure
  Device-related death within 48 hours of the procedure Major bleeding within 48 hours of the procedure
  Device-related AEs within 48 hours, including:
  * Clinical deterioration
  * Pulmonary vascular injury
  * Cardiac injury

CONTACTS AND LOCATIONS:
Overall Officials: Aadi Chachad, Study Director — Sponsor GmbH
Locations (23):
- United States (18):
  - Hartford Hospital, Hartford, Connecticut
  - Ascension Sacred Heart, Pensacola, Florida
  - Emory University, Atlanta, Georgia
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford St John, Detroit, Michigan
  - NYU Langone Health, New York, New York
  - Northwell Health, Staten Island, New York
  - Westchester Medical Center, Valhalla, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Wake Forest Medical Center, Winston-Salem, North Carolina
  - Penn Presbyterian, Philadelphia, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - St Clair Health, Pittsburgh, Pennsylvania
  - MUSC, Charleston, South Carolina
  - Turkey Creek Medical Center, Knoxville, Tennessee
  - Baylor Scott & White, Plano, Texas
  - Carilion, Roanoke, Virginia
- Medical University of Vienna, Vienna, Austria
- Poland (3):
  - St. John Paul II Hospital, Krakow
  - European Health Center Otwock, Otwock
  - Medical University of Warsaw, Warsaw
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No